CLINICAL TRIAL: NCT01542892
Title: Efficacy of Nutritional Supplementation on Physical-activity Mediated Changes in Physical Functioning Older Adults at Risk for Mobility Disability (The VIVE2 Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Uppsala University (Other); Karolinska Institutet (Other); Nestec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10.27.CLI
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Nutrition; Vitamin D; Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supplement (Experimental)
  Interventions: Dietary Supplement: Supplement Intervention
- Placebo (Sham Comparator)
  Interventions: Dietary Supplement: Supplement Intervention
- Exercise (Experimental)
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Participants will complete exercise sessions 3 times per week for 6 months. The exercise sessions will involve walking, lower extremity strength exercises, flexibility, and balance training.
  Arms: Exercise
Dietary Supplement: Supplement Intervention — Participants will be randomly assigned to receive either the nutritional supplement or placebo. The participants will consume on beverage immediately after each exercise session.
  Arms: Placebo; Supplement

SUMMARY:
Several trials have found that nutritional supplementation can elicit an increased rate of skeletal muscle protein synthesis following a single bout of exercise in both young and older individuals. However, there have been no studies that have investigated if nutritional supplementation and exercise can cause a sustained increase in physical functioning and fat free mass, particularly in older adults with functional limitations. This study will compare the effects of a nutritional supplement versus a placebo on exercise training induced changes in physical functioning older adults who are at risk for mobility disability.

DETAILED DESCRIPTION:
Exercise Intervention: Participants will complete exercise sessions 3 times per week for 6 months. The exercise sessions will involve walking, lower extremity strength exercises, flexibility, and balance training.

Supplement Intervention: Participants will be randomly assigned to receive either the nutritional supplement or placebo. The participants will consume on beverage immediately after each exercise session.

Primary Outcome: The primary outcome will be the time to walk 400 meters, expressed as average gait speed during the 400 M walk. All participants must be able to walk 400 meters in <15 minutes at walking at their normal speed. The 400 M walk will be assessed at baseline, 3-months, and 6-months, with the changes at 6-months being the primary outcome.

Secondary Outcome Measures:

* Stair Climb Test
* Body Composition
* Skeletal muscle cross sectional area
* Isokinetic/Isometric peak torque/power
* Hand-grip strength
* Nutritional status
* Quality of Life/Depressive symptoms Expected enrollment: 150 (80 at Tufts University (Boston, MA, USA), 70 at University of Uppsala (Uppsala, Sweden))

ELIGIBILITY:
Inclusion Criteria:

1. Male & Female ≥ 70 yrs
2. Community dwelling
3. Short Physical Performance Battery ≤ 9
4. Willingness to be randomized and come to the laboratory for 6 months
5. Body Mass Index < 35
6. Mini-Mental State Examination >=24
7. Serum 25 (OH) D (22.5 -50 nmol/l)
8. Having obtained his/her informed consent
9. Able to complete 400 M walk within 15 minutes

Exclusion Criteria:

* • Acute or terminal illness; terminal illness with life expectancy less than 12 months, as determined by a physician

  * Current regular use (> 1 per week) of high protein oral nutritional supplements (eg: Boost, Exceed etc…)
  * Current use of Vitamin D supplements, >800 IU/day
  * Myocardial infarction in previous 6 months, symptomatic coronary artery disease, or congestive heart failure.
  * Upper or lower extremity fracture in previous 6 months.
  * Hemoglobin < 10 g/dL, Estimated GFR < 30 mL/min/1.73 m2
  * Uncontrolled hypertension (>150/90 mm Hg).
  * Neuromuscular diseases and drugs which affect neuromuscular function; severe progressive, degenerative neurologic disease
  * Hormone replacement therapy
  * Insulin-dependent diabetes mellitus
  * Milk protein allergy
  * Major surgery in the past 6 months (requiring general anesthesia)
  * Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar, schizophrenia)
  * Excessive alcohol use (>14 drinks per wk)
  * Participation in moderate intensity physical activity > 20 minutes/week
  * Inability to communicate due to severe, uncorrectable hearing loss or speech disorder
  * Severe visual impairment (if it precludes completion of assessments and/or intervention)
  * Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease; wheelchair bound
  * Cancer requiring treatment in the past three years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
  * Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen
  * Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
  * Patient who cannot be expected to comply with treatment, as decided by the Principal Investigator and study physician.
  * Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the clinical site Principal Investigator and/or study physician.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to Walk 400 meters | 6-Month
  The primary outcome will be the time to walk 400 meters, expressed as average gait speed during the 400 M walk. All participants must be able to walk 400 meters in <15 minutes at walking at their normal speed. The 400 M walk will be assessed at baseline, 3-months, and 6-months, with the changes at 6-months being the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Fielding, PhD, Principal Investigator — Tufts University
Locations (2):
- Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Derived] von Berens A, Fielding RA, Gustafsson T, Kirn D, Laussen J, Nydahl M, Reid K, Travison TG, Zhu H, Cederholm T, Koochek A. Effect of exercise and nutritional supplementation on health-related quality of life and mood in older adults: the VIVE2 randomized controlled trial. BMC Geriatr. 2018 Nov 21;18(1):286. doi: 10.1186/s12877-018-0976-z. PMID 30463527
- [Derived] Englund DA, Kirn DR, Koochek A, Zhu H, Travison TG, Reid KF, von Berens A, Melin M, Cederholm T, Gustafsson T, Fielding RA. Nutritional Supplementation With Physical Activity Improves Muscle Composition in Mobility-Limited Older Adults, The VIVE2 Study: A Randomized, Double-Blind, Placebo-Controlled Trial. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):95-101. doi: 10.1093/gerona/glx141. PMID 28977347